CLINICAL TRIAL: NCT06502262
Title: A Comparative Study of Intrathecal Dexmedetomidine and Fentanyl As Additives to Bupivacaine in Pott's Fracture
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MS 571/2023
Record Dates: First submitted 2024-06-22; First posted 2024-07-16 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-02

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Fentanyl; Dexmedetomidine

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- • control (Active Comparator): • Drug: hyperbaric bupivacaine this group will be given 3 ml (15mg) of 0.5% hyperbaric bupivacaine+0.5 ml of normal saline intrathecally.
  Interventions: Drug: Bupivacaine Hydrochloride
- •Fentanyl group (Active Comparator): •Drug: Fentanyl this group will be given 3 ml (15 mg) of 0.5% hyperbaric bupivacaine+0.5 ml (25μg) of fentanyl intrathecally.
  Interventions: Drug: Bupivacaine Hydrochloride; Drug: Fentanyl
- •Dexmedetomidine group (Active Comparator): •this group will be given 3 ml (15 mg) of 0.5% hyperbaric bupivacaine+0.5 ml (5μg) of diluted dexmedetomidine intrathecally
  Interventions: Drug: Bupivacaine Hydrochloride; Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride — patient will be given 3ml (15mg) of 0.5% hyperbaric bupivacaine + 0.5 ml of normal saline intrathecally.
Drug: Fentanyl — patients will be given 3ml (15mg) of 0.5%hyperbaric bupivacaine +0.5ml (25 microgram) of fentanyl intrathecally
  Arms: •Fentanyl group
Drug: Dexmedetomidine — patient will receive 3ml (15mg) of .05 hyperbaric bupivacaine 0.5ml(5 microgram) of diluted dexmedetomidine intrathecally
  Other Names: precedex
  Arms: •Dexmedetomidine group

SUMMARY:
The aim of this study is to compare the addition of intrathecal dexmedetomidine or fentanyl as adjuvants to hyperbaric bupivacaine in the onset and duration of sensory and motor block, and postoperative analgesia.

DETAILED DESCRIPTION:
The aim of this study is to compare the addition of intrathecal dexmedetomidine or fentanyl as adjuvants to hyperbaric bupivacaine in the onset and duration of sensory and motor block, and postoperative analgesia. All patients will be assessed preoperatively by careful history taking, full physical examination, and laboratory evaluation. An informed written consent will be taken from every patient just before the surgery. On arrival to the operating room, baseline parameters such as ECG, mean arterial blood pressure, heart rate, and oxygen saturation will be recorded. Intravenous line will be inserted and IV Ringer's solution will be started, 500ml bolus will be given as a preload over 20 min before performing spinal anesthesia and maintenance volume of 10ml\kg.

For each group, patients will be put in sitting position, lumbar puncture will be performed under complete aseptic precautions, local anesthesia will be administered by infiltration of the skin and subcutaneous tissues with 3-5 ml lidocaine 1% at L3-L4 and A 25-G needle will be used.

* Group 1: (Control group) (20 cases): patients will receive 3 ml (15mg) of 0.5% hyperbaric bupivacaine+0.5 ml of normal saline intrathecally.
* Group 2: (Fentanyl group) (20 cases): patients will receive 3 ml (15 mg) of 0.5% hyperbaric bupivacaine+0.5 ml (25μg) of fentanyl intrathecally.
* Group 3: (Dexmedetomidine group) (20 cases): patients will receive 3 ml (15 mg) of 0.5% hyperbaric bupivacaine+0.5 ml (5μg) of diluted dexmedetomidine intrathecally.

ELIGIBILITY:
Inclusion Criteria:

* • ASA I or ASA II patients Scheduled for pott's, of either sex.

  * Age 21-55 years.
  * Height 160 to 190 cm.
  * BMI ≤40.
  * Procedure duration ≤ 90 minutes

Exclusion Criteria:

* • Patients with known neurologic and psychiatric illness.

  * Contraindications for spinal anesthesia as patient refusal, bleeding or coagulation test abnormalities, local skin infection at spinal lumbar region, raised intracranial pressure and hypovolemia.
  * Spine abnormalities.
  * Systemic disorders like hematological, respiratory, cardiac, renal or hepatic insufficiency.
  * Allergy to any of the drugs used in the study.
  * Women with pregnancy and lactation

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
motor blockade onset | from injection up to Modified Bromage score 1 ( 5 minutes)
  Onset of motor block (defined as time in minutes from the end of drug injection intrathecally until patient is unable to move the hip, knee, and ankle)
sesnory onset | from injection up to s1 regression ( 5 minutes)
  defined as time in minutes to reach highest sensory level) will be tested every minute after intrathecal injection until it reach the highest level. It will be assessed by pin prick and cold application
post operative analgesia | from injection up to 24 hours post operative
  will be evaluated using a visual analog scale (VAS),

SECONDARY OUTCOMES:
drop in mean blood pressure | from injection up to 24 hours post operative
  using non invasive arterial blood pressure monitoring
drop in oxygen saturation | from injection up to24hours post operative
  using pulse oximiter
drop in heart rate | from injection up to 24 hours post operative
  using ecg monitoring

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Abbassia, Egypt

IPD SHARING:
Plan to Share IPD: No